CLINICAL TRIAL: NCT06921317
Title: Proof of Concept Clinical Trial of Gene Therapy GVB-2001 Delivered Via Intracameral Injection for the Treatment of Primary Open Angle Glaucoma
Brief Title: GVB-2001 Gene Therapy Via Intracameral Injection for the Treatment of Primary Open Angle Glaucoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IVIEW Therapeutics Inc. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GVB-2001-GLU-IIT
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Primary Open-Angle Glaucoma (POAG)
Keywords: glaucoma; gene therapy; rho gene; trabecular meshwork; dnRhoA; IOP reduction; AAV; scAAV
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Night Blindness, Congenital Stationary, Autosomal Dominant 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: POAG patient without vision (Experimental): Low dose or high dose GVB-2001 25ul will be injected once into the anterior chamber by the investigator at visit 2.
  Interventions: Drug: GVB-2001-high dose; Drug: GVB-2001-low dose
- Group 2: POAG patient with vision (Experimental): Low dose or high dose GVB-2001 will be injected once into the anterior chamber by the investigator at visit 2.
  Interventions: Drug: GVB-2001-high dose; Drug: GVB-2001-low dose

INTERVENTIONS:
Drug: GVB-2001-high dose — GVB-2001 is a self-complementary adeno-associated viral vector (scAAV) injection to deliver human dnRhoA gene to trabecular meshwork cells in patients with primary open angle glaucoma. A single dose of high dose GVB-2001 will be injected intracamerally to the target interventional eye.
Drug: GVB-2001-low dose — GVB-2001 is a self-complementary adeno-associated viral vector (scAAV) injection to deliver human dnRhoA gene to trabecular meshwork cells in patients with primary open angle glaucoma. A single dose of low dose GVB-2001 will be injected intracamerally to the target interventional eye.

SUMMARY:
This is an investigator initiated, single center, open label, non-randomized, exploratory clinical study. The purpose is to assess the safety and preliminary efficacy of gene therapy GVB-2001 (ScAAV2-dnRhoA) delivered via intracameral injection to the anterior segment of the eye for the treatment of subjects with primary open-angle glaucoma. At least 12 primary open angle glaucoma (POAG) patients with high intraocular pressure (IOP) will be divided into two experimental groups. Each experimental group will receive either a low dose or a high dose interacameral injection of GVB-2001. The optimal dose will be selected based on the trial results for future development of GVB-2001.

Safety Review Committee, SRC will be set up for safety assessment of the study. The study subjects included will be 18 to 65 years of age (inclusion) and are diagnosed with primary open-angle glaucoma (POAG) for 1 year or more. Only participants who provide informed consent prior to all screening procedures will be eligible for enrollment into the trial.

DETAILED DESCRIPTION:
This research plans to recruit at least 12 high intraocular pressure of primary open-angle glaucoma (POAG) patients in one clinical center and divide into two groups. Six primary glaucoma (POAG) patients with elevated intraocular pressure and no vision in the target eye will be enrolled in trial group 1. They will be divided into two dose groups: low-dose group (n = 3) and high-dose group (n = 3). The safety review committee (SRC) will determine whether to enter the high- dose group after the last subject in the low-dose group has completed the Dose limited toxicity (DLT) assessment. In group 2, 6 primary open-angle (POAG) patients with normal visual acuity and high intraocular pressure will be enrolled. The patients will be divided into low-dose group (3 subjects) and high-dose group (3 subjects). The safety review committee (SRC) will determine whether to enter the low-dose group of trial group 2, and whether to enter the high-dose group of trial group 2, after the completion of the evaluation of DLT in the low-dose group of trial group 1. During the study of trial group 2, the safety review committee (SRC) will determine whether to add another optimized dose group to trial group 2, and determine the optimized therapeutic dose and the number of subjects in the optimized dose group.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects volunteered to participate in the clinical study and signed written informed consent;
2. Aged 18 to 70 years old (inclusive), men and women;
3. Primary open angle glaucoma (POAG) with a history of diagnosis ≥1 year;
4. Participants in good general health and have no clinically significant systemic disease, as determined by medical history, physical examination, and screening laboratory evaluation.
5. To comply with the requirements, willing to accept all the diagnosis and treatment plan, laboratory tests and other specified testing, etc.;
6. Consent is obtained for an extended safety visit after 1 year.

Special eligibility criteria for trial group 1:

1. no vision in the target eye;
2. The intraocular pressure (IOP) of the target eye was ≤40mmHg and > 21 mmHg after combined treatment with 2 or more IOP-lowering drugs.

Special inclusion criteria for trial group 2:

1. The intraocular pressure (IOP) of the target intervention eye was no more than 30mmHg, and the IOP was more than 21 mmHg after receiving combination therapy of 2 or more IOP-lowering drugs;
2. The Shaffer gonioscopy scores of the target intervention eyes were all greater than 3.
3. The best corrected distance visual acuity of the target intervention eyes was at least 0.8 (logMAR4.9) and above.

Exclusion Criteria:

1. Secondary glaucoma;
2. Any active or recurrent intraocular infection or inflammation, including but not limited to uveitis;
3. Severe dry eye or clinically significant active keratopathy in the target eye;
4. No intraocular pressure measurement was performed under any circumstances;
5. Allergies to drugs or their excipient to be used in clinical studies;
6. Ocular trauma in either eye within 6 months before screening, or eye surgery or nonrefractive laser therapy within 3 months before screening;
7. A clinically significant history of herpes simplex or herpes zoster keratitis;
8. A positive test for hepatitis B virus (HBV) HBsAg or HBV-DNA, hepatitis C virus (HCV) HCAb, or Epstein-Barr virus, or cytomegalovirus (CMV);
9. Syphilis antibody and HIV antibody were positive.
10. Severe active systemic bacterial, viral, fungal, malaria, or parasitic infections;
11. Any past or present malignant tumor, myeloproliferative disorder or immunodeficiency disease;
12. May interfere with the clinical significance of this study of systemic disease (including, active hepatitis, liver cirrhosis, liver fibrosis uncontrolled hypertension, myocardial infarction and myocarditis, arrhythmia, stroke, acute or chronic renal insufficiency, uncontrolled endocrine system diseases such as diabetes, thyroid function hyperfunction, Severe pulmonary hypertension, chronic obstructive pulmonary disease (copd), interstitial pneumonia, etc.);
13. Any serious mental illness;
14. Have participated in other clinical trials and received a medication or medical device intervention within 1 month before screening;
15. And women of childbearing age who are pregnant, breastfeeding, planning to become pregnant, or who are not using a medically acceptable form of birth control. Excludes women of childbearing age who have been sterilized for 1 year after menopause or 3 months after surgery;
16. Other subjects judged by the clinical investigator to be ineligible for inclusion.

Special Exclusion Criteria for trial group 1:

1) The serum Anti-AAV2 neutralizing antibody titer was > 1:200 at the time of screening.

Special Exclusion Criteria for trial group 2:

1. Retinal diseases that might have interfering with the study: quadrantinal blindness of unknown cause, wet age-related macular degeneration, retinal vein occlusion, cystoid macular edema, macular hole, maculopathy with neovascularization, and central serous retinopathy;
2. Narrow anterior chamber Angle, congenital Angle closure glaucoma or room, clinically significant peripheral anterior chamber adhesion or anterior chamber Angle surgery/laser treatment cause extensive catarrhal adhesion of history;
3. The central corneal thickness was less than 480μm or more than 620μm.
4. Presence of severe visual field impairment (e.g., mean deviation less than -12 dB or mean visual field defect greater than 2 dB/ year, as assessed by a perimetry analyzer)
5. The target eye had undergone intraocular anti-glaucoma surgery or anti- glaucoma laser surgery;
6. The serum Anti-AAV2 neutralizing antibody titer was > 1:600 at the time of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The number and proportion of subjects with IOP ≤21mmHg | Day 28, Day 60, Day 90, 6-Month, and 12-Month after GVB-2001 administration.
The number and proportion of subjects whose IOP decreased by ≥20% from baseline | Day 28, Day 60, Day 90, 6-Month, and 12-Month after GVB-2001 administration.
Ocular adverse events (AEs) : the characteristics of AES, including endophthalmitis, eyelid edema, and corneal injection site reaction | Day 1, Day 3, Day 7, Day 14, Day 28, Day 60, Day 90, 6-Month and 12--Month after GVB-2001 administration.

SECONDARY OUTCOMES:
Type, number, and incidence of systemic adverse events and serious adverse events | Adverse events (AEs): The type, number and incidence of AEs and serious adverse events (SAEs) will be analysized within 12 months after GVB-2001 administration.
The number of ocular malignancies related to GVB-2001 injection occurred after treatment | After GVB-2001 Administration up to 5 years.
RhoA protein concentration in blood | Day 7, Day 28, and 12-Month after GVB-2001 administration
RhoA protein concentration in urine | Day 7, Day 28, and 12-Month after GVB-2001 administration
RhoA protein concentration in tears | Day 7, Day 28, and 12-Month after GVB-2001 administration
AAV2 Virus Shedding in blood | Day 7, Day 28, and Month 12 after GVB-2001 administration
AAV2 Virus Shedding in urine | Day 7, Day 28, and 12-Month after GVB-2001 administration
AAV2 Virus Shedding in tears | Day 7, Day 28, and 12-Month after GVB-2001 administration
Humoral immunity response | Day 7, Day 28, and 12-Month after GVB-2001 administration
  Humoral immunity response is evaluated by comprehensive judgements of IgG, IgM, IgA, complements and Light chains in blood. It's applied to assess safety.
Cellular immunity response | Day 7, Day 28, and 12-Month after GVB-2001 administration
  Cellular immunity response is evaluated by comprehensive judgements of CD3 CD4 CD8 in blood. It's applied to assess safety.
AAV2 antibody titer level in blood | Day 7, Day 28, and 12-Month after GVB-2001 administration.
  Compare antibody level to baseline. It's applied to assess safety.
Occurance of Dose limiting toxicity (DLT) as determined by the Safety Monitoring Committee (SRC) | Day 28 after GVB-2001 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Lu, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No